CLINICAL TRIAL: NCT04581005
Title: Prehabilitation to Enhance Functional Capacity in Esophageal Cancer Care
Brief Title: Prehabilitation in Esophageal Cancer Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Franco Carli, Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MUHC 2019-5387
Record Dates: First submitted 2020-08-15; First posted 2020-10-09 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Preoperative Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervised Prehabilitation (Experimental): Prehabilitation will include exercise, nutrition, and anxiety-coping intervention.
  This group will receive a supervised, in-hospital training.
  Interventions: Behavioral: Prehabilitation
- Home-based Prehabilitation (Experimental): Prehabilitation will include exercise, nutrition, and anxiety-coping intervention.
  This group will receive a home-based training.
  Interventions: Behavioral: Prehabilitation

INTERVENTIONS:
Behavioral: Prehabilitation — Endurance and Resistance Exercise, Nutrition therapy, reducing intervention during the whole preoperative period

SUMMARY:
Prehabilitation utilizes the preoperative period to prevent or attenuate the treatment-related functional decline and its consequences. This project aims at testing feasibility and effectiveness of multimodal prehabilitation in esophageal cancer care.

DETAILED DESCRIPTION:
While evidence on prehabilitation is mounting, upper gastrointestinal surgery still remains under-investigated. This trial aims to explore the effect of prehabilitation over the whole perioperative trajectory, including neo-adjuvant treatment (NAT).

Multimodal prehabilitation includes exercise, nutrition therapy, and mental distress coping strategies. In the context of a multimodal approach, the two groups follow different exercise prescriptions: high-intensity interval supervised training prescribed accordingly cardiopulmonary exercise testing (CPET)-derived variables, versus a home-based program. For both groups, multimodal prehabilitation is prescribed over the whole preoperative period, including during NAT.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-metastatic esophageal cancer undergoing neo-adjuvant chemotherapy and surgery.

Exclusion Criteria:

* co-morbid medical, physical and mental conditions that contraindicate exercise or oral nutrition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2019-08-19 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Oxygen consumption (VO2) | Change from baseline to 2 months after surgery
  Oxygen consumption at anaerobic threshold (VO2 at AT) measured with cardiopulmonary exercise testing (CPET)
Oxygen consumption (VO2) | Change from baseline to post neo-adjuvant therapy (average duration 6-8 weeks)
  Oxygen consumption at anaerobic threshold (VO2 at AT) measured with cardiopulmonary exercise testing (CPET)

CONTACTS AND LOCATIONS:
Overall Officials: Enrico M Minnella, MD PhD, Principal Investigator — McGill University
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No